CLINICAL TRIAL: NCT02866825
Title: A Phase II Randomized, Placebo-controlled, Double-blind, Dose-escalation Study to Evaluate Safety, Pharmacokinetics and Pharmacodynamic Dose Response Relationship of IFX-1 in Patients Undergoing Complex Cardiac Surgery
Brief Title: Studying Complement Inhibition in Complex Cardiac Surgery
Acronym: CARDIAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: InflaRx GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IFX-1-P2.2; 2015-003036-12 (EudraCT Number)
Record Dates: First submitted 2016-06-17; First posted 2016-08-15 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Systemic Inflammatory Response Syndrome; C.Surgical Procedure; Cardiac
Keywords: Inflammation; Systemic Inflammatory Response Syndrome; Pathologic Processes; Organ Dysfunction
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Inflammation; Pathologic Processes | interventions — vilobelimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IFX-1 (Active Comparator): dose escalating single i.v. administration of IFX-1 (verum)
  Interventions: Biological: IFX-1
- Placebo (Placebo Comparator): dose escalating mimicing single i.v. administration of placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: IFX-1
  Arms: IFX-1
Biological: Placebo
  Arms: Placebo

SUMMARY:
The trial enrolls patients undergoing a complex cardiac surgery. The primary goal of the trial is to evaluate the pharmacodynamic dose response relationship of the monoclonal antibody IFX-1 in these patients. In addition, this trial further aims to characterize the safety and the pharmacokinetics of IFX-1 as well as to collect first data on its efficacy on clinical surrogate endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years old
2. Written informed consent
3. One of the following cardiac surgical procedures is planned with Cardiopulmonary bypass (CPB):

   * Single valve surgery in combination with at least two coronary artery bypass grafts (CABGs)
   * Multiple valve surgery with or without CABG
   * Single or multiple valve surgery in combination with ascending aorta procedure with or without additional CABG
   * Re-surgery of aortic valve, mitral valve, aortic arch or ascending aorta with or without CABG
4. Cardiac surgery is performed electively

Exclusion Criteria:

1. Weight > 130 kg
2. The following cardiac surgical procedures:

   * Cardiac surgical procedure is planned as minimally invasive procedure (e.g., without thoracotomy or with lateral incision, minimal thoracotomy)
   * Cardiac surgery with an expected CPB time less than 100 minutes
3. Other cardiac and vascular diseases and/or procedures:

   * Prior cardiac surgery within the past 6 months
   * History of heart transplantation or planned heart transplantation
   * Requiring inotropic, vasopressor or mechanical circulatory support
   * Requiring ventilatory support
4. Other disease or condition that is likely to interfere with the evaluation of the study drug:

   * Active infective endocarditis
   * Stroke or transient ischemic attack (TIA) within the last 6 months
   * Concomitant disease with a life expectancy of less than 6 months
   * Cardiopulmonary resuscitation within the last 4 weeks
   * Patients requiring renal replacement therapy
5. Cerebrovascular disease requiring concomitant carotid endarterectomy
6. Active infection with or without a temperature greater than 38°C
7. Presence of systemic inflammatory response syndrome defined as occurrence of at least 2 out of the following 4 criteria:

   * Fever > 38.0°C or hypothermia < 36.0°C
   * Tachycardia > 90 beats/minute
   * Tachypnea > 20 breaths/minute
   * Leucocytosis > 12 x 109/l or leucopenia < 4 x 109/l or > 10% immature neutrophils (bands)
8. Positive test for human immunodeficiency virus (HIV), hepatitis B or C
9. One of the following abnormal laboratory results:

   * Hemoglobin < 5 mmol/l (< 8.06 g/dl)
   * Total bilirubin ≥ 2 x upper normal limit (UNL)
   * CRP > 3 x UNL
   * ALAT > 3 x UNL
   * ASAT > 3 x UNL
   * White blood cell count < 2,500/mm³
   * White blood cell count > 12,000/mm³
10. Prohibited concomitant medications:

    * Immunomodulatory drugs within past 30 days (e.g., TNF-inhibitors)
    * Immunosuppressive drugs within past 30 days (e.g., cyclosporine, tacrolimus)
    * High dose corticosteroids (e.g., > 50 mg prednisone/day or equivalent) within past 14 days
    * Any systemic anticancer treatment within the past 3 months
11. Planned corticosteroid pulse therapy to prevent SIRS
12. Patients with known hypersensitivity to any constituent of the investigational medicinal product (IMP)
13. General exclusion criteria:

    * Pregnant (in women of childbearing potential an urine pregnancy test has to be performed) or breast-feeding women
    * Women with childbearing potential (defined as within two years of their last menstruation) not willing to practice appropriate contraceptive measures (e.g., implanon, injections, oral contraceptives, intrauterine devices, partner with vasectomy, abstinence) while participating in the trial
    * Participation in any interventional clinical trial within the last three months
    * Prior randomization in this clinical trial (screen failures can be re-screened, if appropriate)
    * Alcohol, drug, or medication abuse
    * Employee at the study site, spouse/partner or relative of any study staff (e.g., investigator, sub-investigators, or study nurse) or relationship to the sponsor
    * No commitment to full aggressive life support (e.g., DNR order)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2016-05; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Peak level of IL-6 | From prior study drug administration until 24h after start of cardiopulmonary bypass (CPB) (CPB)

SECONDARY OUTCOMES:
Plasma concentration of IFX-1 at each timepoint measured | Data will be collected at the following approximate time points: prior study drug administration; 30 min after start of infusion; up to 10 min after cessation of CPB; 3h, 12h, 24h, 48h, 96h, and 168h after start of CPB; Day 15
Maximum observed concentration (Cmax) of IFX-1 | Data will be collected at the following approximate time points: prior study drug administration; 30 min after start of infusion; up to 10 min after cessation of CPB; 3h, 12h, 24h, 48h, 96h, and 168h after start of CPB; Day 15
Area under the curve (AUC) of plasma concentration of IFX-1 | Data will be collected at the following approximate time points: prior study drug administration; 30 min after start of infusion; up to 10 min after cessation of CPB; 3h, 12h, 24h, 48h, 96h, and 168h after start of CPB; Day 15
Plasma concentration of free, detectable C5a at each timepoint measured | Data will be collected at the following approximate time points: prior study drug administration, prior start of CPB, up to 10 min after cessation of CPB; 3h, 6h, 12h, 24h, 48h, 96h, and 168h after start of CPB; Day 15
Serum levels of CH50 at each timepoint measured | Data will be collected at the following approximate time points: prior study drug administration, prior start of CPB, up to 10 min after cessation of CPB; 3h, 6h, 12h, 24h, 48h, 96h, and 168h after start of CPB; Day 15
Serum levels of IL-6 compared to baseline | Data will be collected at the following approximate time points: prior study drug administration, up to 10 min after cessation of CPB; 3h, 6h, 12h, 24h, 48h, and 96h after start of CPB; Day 15
Serum levels of IL-8 compared to baseline | Data will be collected at the following approximate time points: prior study drug administration, up to 10 min after cessation of CPB; 3h, 6h, 12h, 24h, 48h, and 96h after start of CPB; Day 15
Incidence of patients with Adverse Events (AEs) and Serious Adverse Events (SAEs) until Day 29 | From screening visit until Day 29
Number of patients with detection of anti-drug-antibodies | Up to Day 15
Number of patients that are successfully extubated 24h after end of surgery | 24h after end of surgery
Number of patients with consecutive invasive ventilation for more than 48h after end of surgery | 48h after end of surgery
Number of patients that are weaned of any vasopressor use 24h after end of surgery | 24h after end of surgery
Number of patients with SIRS 24h, 48h and 96h after start of CPB | 24h, 48h and 96h after start of CPB

CONTACTS AND LOCATIONS:
Overall Officials: Torsten Doenst, Prof. Dr., Principal Investigator — University Hospital Jena
Locations (10):
- Germany (10):
  - Study Site, Aachen
  - Study Site, Dortmund
  - Study Site, Dresden
  - Study Site, Freiburg im Breisgau
  - Study Site, Heidelberg
  - Study Site, Jena
  - Study Site, Kiel
  - Study Site, Leipzig
  - Study Site, Trier
  - Study Site, Tübingen

IPD SHARING:
Plan to Share IPD: No